CLINICAL TRIAL: NCT04438239
Title: Rehabilitation Needs After COVID-19 Hospital Treatment (REACT): an Observational Study
Brief Title: Rehabilitation Needs After COVID-19 Hospital Treatment
Acronym: REACT
Status: Completed | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: 428/2020/OSS/AUSLRE
Record Dates: First submitted 2020-06-10; First posted 2020-06-18 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Covid-19
Keywords: Covid-19; Rehabilitation; patients' needs
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covid-19 discharged: Patients affected by COVID-19 and discharged from hospital wards of the Azienda USL- IRCCS Of Reggio Emilia (Italy).
  Interventions: Other: none, this study is observational

INTERVENTIONS:
Other: none, this study is observational — none, this study is observational

SUMMARY:
The onset of Coronavirus Disease 2019 (COVID-19) in the first months of 2020 had a huge impact on Italian population and Healthcare System, with more than 150.000 total confirmed cases1. SARS-CoV-2 is a highly contagious new virus, causing an influenza like illness and respiratory tract infection demonstrating fever (89%), cough (68%), fatigue (38%), sputum production (34%) and/or shortness of breath (19%).

The aim of this observational study is to detect symptoms, disabilities, participation and the lived experience of the disease in individuals affected by COVID-19 two months after the hospital discharge.

DETAILED DESCRIPTION:
The onset of Coronavirus Disease 2019 (COVID-19) in the first months of 2020 had a huge impact on Italian population and Healthcare System, with more than 150.000 total confirmed cases. SARS-CoV-2 is a highly contagious new virus, causing an influenza like illness and respiratory tract infection demonstrating fever (89%), cough (68%), fatigue (38%), sputum production (34%) and/or shortness of breath (19%). The spectrum of disease severity ranges from an asymptomatic infection or mild upper respiratory tract illness (80% of cases), to 15% of cases with severe infection with fever, cough, fatigue and shortness of breath, requiring oxygen, and 5% are severe viral pneumonia with respiratory failure requiring ventilation and life support and/or death. At present, clinicians do not know the real impact of Coronavirus Disease on patients' performances, functional status and QoL. Patients admitted to hospital experience fever, cough, dyspnea, muscle soreness and/or acute respiratory distress syndrome but healthcare professionals observe also anxiety, depression and important functional limitations during hospital stay. This situation is expected to have a significant negative impact in the short term, mainly for patients affected by other medical conditions and it may lead to deconditioning, fatigue, isolation, poor functional status and QoL.

In the first months after COVID-19 outbreak, researchers focused their studies on infection epidemiology, transmission, COVID-19 diagnosis and medical treatments. As the epidemic progresses, a large part of patients is expected to come out of the acute phase, and they may need adequate rehabilitation to face functional limitations and return to previous levels of participation.

To date, the very few studies published on the rehabilitation of positive and symptomatic patients with COVID-19 focused on pulmonary rehabilitation guidelines or on implications for rehabilitation services. To our knowledge, no clinical trial on rehabilitation intervention for patients after COVID-19 is ongoing. Our research group set up an observational study to detect patients' rehabilitation needs after COVID-19, collecting data on symptoms, impairments, functional abilities and participations to social life in the first months after hospital discharge.

The aim of this observational study is to detect symptoms, disabilities, participation and the lived experience of the disease in individuals affected by COVID-19 two months after the hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* age>18,
* positive at COVID-19
* manifesting symptoms that required hospitalization, that is history of fever or pneumonia or other symptoms COVID-19 related.

Exclusion Criteria:

* asymptomatic individuals COVID-19 positive that were hospitalized for reasons other than COVID-19;
* dementia;
* psychiatric disorders
* other diseases preventing people to participate to the rehabilitation assessments provided by this protocol;
* acute or post-acute clinical conditions causing disability itself (e.g.: major neurological disease, such as recent stroke, TBI, etc., or recent surgical intervention, or heart failure, etc.),
* previous complete dependence in ADLs .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients hospitalized for COVID-19 and discharged from hospital wards of the Azienda USL- IRCCS Of Reggio Emilia (Italy) from April to June 2020
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
number of participants with considerable dyspnea: Medical Research Council (MRC, 0-4, lower score better outcome) | 2-months after hospital discharge
  Dyspnea will be measured with Medical Research Council (MRC), minimum value 0-maximum value 4, lower value= better outcome
number of participants with fatigue | 2-months after hospital discharge
  Fatigue will be assessed with Fatigue Severity Scale (FSS), minimum value 9-maximum value 63, lower value=better outcome
number of participants with anxiety | 2-months after hospital discharge
  anxiety will be assessed with Hospital Anxiety and Depression Scale (HADS), subscale 'Anxiety', minimum value 0-maximum value 24, lower score=better outcome, cut-off for clinically significant anxiety score>7
number of participants with depression | 2-months after hospital discharge
  depression will be assessed with Hospital Anxiety and Depression Scale (HADS), subscale 'Depression', minimum value 0-maximum value 24, lower score=better outcome, cut-off for clinically significant depression score>7

SECONDARY OUTCOMES:
level of independence in B-ADL | 2-months after hospital discharge
  independence or disability will be assessed with Barthel Index (BI), minimum score 0- maximum score 100, higher score=better outcome
level of participation in social | 2-months after hospital discharge
  reintegration into normal social activities (e.g. recreation, movement in the community, and interaction in family or other relationships) will be assessed with Reintegration to Normal Living Index (RNLI), minimum score 0-maximum score 100, higher score=better outcome
description of qualitative data about patients' experience | 2-months after hospital discharge
  open ended questions will be recorded, transcribed verbatim and analyzed (two questions addressed to symptoms and limitations in activities that patients may have experienced during hospitalization or after discharge)

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Fugazzaro, MD, Principal Investigator — Azienda USL - IRCCS of Reggio Emilia (Italy)
Locations (1):
- Azienda USL-IRCCS S.Maria Nuova Hospital, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boldrini P, Bernetti A, Fiore P; SIMFER Executive Committee, SIMFER Committee for International Affairs. Impact of COVID-19 outbreak on rehabilitation services and Physical and Rehabilitation Medicine physicians' activities in Italy. An official document of the Italian PRM Society (SIMFER). Eur J Phys Rehabil Med. 2020 Jun;56(3):316-318. doi: 10.23736/S1973-9087.20.06256-5. Epub 2020 Mar 16. No abstract available. PMID 32175719
- [Derived] Fugazzaro S, Denti M, Mainini C, Accogli MA, Bedogni G, Ghizzoni D, Bertolini A, Esseroukh O, Gualdi C, Schiavi M, Braglia L, Costi S. Sex differences and rehabilitation needs after hospital discharge for COVID-19: an Italian cross-sectional study. BMJ Open. 2022 May 18;12(5):e055308. doi: 10.1136/bmjopen-2021-055308. PMID 35584875
- [Derived] Schiavi M, Fugazzaro S, Bertolini A, Denti M, Mainini C, Accogli MA, Bedogni G, Ghizzoni D, Esseroukh O, Gualdi C, Costi S. "Like before, but not exactly": the Qualy-REACT qualitative inquiry into the lived experience of long COVID. BMC Public Health. 2022 Mar 28;22(1):599. doi: 10.1186/s12889-022-13035-w. PMID 35346138